CLINICAL TRIAL: NCT05453968
Title: A Phase 3 Study to Evaluate the Safety and Pharmacokinetics of Berotralstat Prophylaxis in Children With Hereditary Angioedema Who Are 2 to < 12 Years of Age
Brief Title: Berotralstat Treatment in Children With Hereditary Angioedema
Acronym: APeX-P
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCX7353-304; 2021-005932-50 (EudraCT Number)
Record Dates: First submitted 2022-06-30; First posted 2022-07-12 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Hereditary Angioedema; Pediatric
Keywords: Berotralstat; BCX7353; Orladeyo®; once a day; Hereditary angioedema (HAE); Pediatric; oral once a day dosing; kallikrein inhibitor
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — berotralstat

STUDY DESIGN:
Intervention Model Description: This is a sequential, three-part, open-label study. Minimum participation in this study is expected to be 24 weeks in the SOC treatment period through Part 1 of the study and up to an additional 132 weeks in Parts 2 and 3.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Berotralstat (Experimental): Berotralstat administered once daily in 4 dose cohorts determined by participant weight. Cohorts 1 and 2 will enroll in parallel. After 4 participants from Cohort 1 and 2, with ≥ 2 subjects from Cohort 2, have reached Week 2, Cohort 3 will open for enrollment. Cohort 4 will open for enrollment, after ≥ 4 subjects in Cohort 3 have reached Week 2. Prior to dosing Cohort 3 and 4, available PK and safety data will be reviewed to confirm it is safe to proceed and the appropriate weight bands for each. BioCryst will notify sites when Cohorts 3 and 4 are open for enrollment.
  Interventions: Drug: Berotralstat

INTERVENTIONS:
Drug: Berotralstat — Administered orally once daily at a weight-based dose in up to 4 cohorts
  Other Names: BCX7353; Orladeyo®

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK) and safety of berotralstat to determine the appropriate weight-based dose for pediatric participants 2 to < 12 years old for prophylactic treatment to prevent attacks of hereditary angioedema (HAE).

DETAILED DESCRIPTION:
This is a single-arm, open-label study designed to evaluate the PK and safety of berotralstat weight-based treatment for the prevention of hereditary angioedema attacks in pediatric participants 2 to < 12 years of age. This study will consist of two treatment periods: a 12-week standard-of-care (SOC) treatment period followed by an open-label berotralstat treatment period lasting up to 144 weeks.

Participants will be enrolled into 4 dose cohorts; participant weight will be used to determine assignment to each cohort with the higher weight cohorts (Cohorts 1 and 2) enrolling first and in parallel. Safety assessments and PK modelling from all available PK data will then be used to confirm the weight bands for sequentially enrolling Cohorts 3 and 4.The effectiveness of berotralstat in this population will be summarized using descriptive statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant, non-lactating females 2 to < 12 years of age
* Body weight ≥ 12 kg
* Clinical diagnosis of HAE
* In the opinion of the investigator, the participant would benefit from long term oral HAE prophylaxis

Exclusion Criteria:

* Concurrent diagnosis of any other type of recurrent angioedema
* Known family history of sudden cardiac death
* Creatinine clearance using the modified Schwartz formula of ≤ 30 mL/min/1.73 m2
* Aspartate aminotransferase or alanine aminotransferase value ≥ 3 × the upper limit of the age-appropriate normal reference range value
* Clinically significant abnormal ECG including but not limited to, a corrected QT interval calculated using Fridericia's correction > 450 msec, or ventricular and/or atrial premature contractions that are more frequent than occasional, and/or as couplets or higher in grouping
* Current participation in any other investigational drug study or received another investigational drug within 30 days of enrollment

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics: Cmax | Predose and multiple timepoints up to 24 hours postdose
  Maximum plasma concentration of berotralstat
Pharmacokinetics: AUC0-tau | Predose and multiple timepoints up to 24 hours postdose
  Area under the plasma concentration berotralstat time curve from time zero to the end of dosing (tau)
Pharmacokinetics: CL/F | Predose and multiple timepoints up to 24 hours postdose
  Apparent oral clearance of berotralstat

SECONDARY OUTCOMES:
Frequency and severity of adverse events (AEs) and serious adverse events (SAEs) | Over 144 weeks
Frequency and severity of hereditary angioedema (HAE) attacks | Over 48 weeks

OTHER OUTCOMES:
Acceptability/palatability of berotralstat oral granules using a self-reported taste rating scale designed with images centered on taste | Time of first dose (Day 1)
  TASTY; 7-point scale [0 "worst" to 6 "best"]

CONTACTS AND LOCATIONS:
Overall Officials: Jolanta Bernatoniene, MD, Principal Investigator — Bristol Royal Hospital for Children
Locations (15):
- Investigative Site #1, Vienna, Austria
- Investigative Site #1, Ottawa, Ontario, Canada
- France (3):
  - Investigative Site #3, Grenoble
  - Investigative Site #2, Marseille
  - Investigative Site #1, Paris
- Germany (2):
  - Investigative Site #1, Berlin
  - Investigative Site #2, Frankfurt
- Israel (2):
  - Investigative Site #2, Haifa
  - Investigative Site #1, Tel Aviv
- Investigative Site #1, Padua, Italy
- Investigative Site #1, Krakow, Poland
- Investigative Site #1, Sângeorgiu de Mureş, Romania
- Spain (2):
  - Investigative Site #1, Madrid
  - Investigative Site #2, Málaga
- Investigative Site #1, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bernatoniene J, Bourgoin-Heck M, Cancian M, Yang W, Hagin D, Pagnier A, Stobiecki M, Kinaciyan T, Phillips-Angles E, Gayet S, Bara NA, Hunter J, Mateescu E, DeSpirito M, Johnston D, Long D, Iocca H, Petroni D, Aygoren-Pursun E. Oral berotralstat for hereditary angioedema prophylaxis in patients aged 2 to <12 years: APeX-P interim results. Ann Allergy Asthma Immunol. 2025 Dec;135(6):681-688.e3. doi: 10.1016/j.anai.2025.07.012. Epub 2025 Jul 25. PMID 40716738